CLINICAL TRIAL: NCT03041662
Title: Surveillance Study for Early Detection of Cholangiocarcinoma (CCA) in Primary Sclerosing Cholangitis (PSC)
Acronym: PSC
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Annika Bergquist, professor, Karolinska University Hospital
Other Study IDs: 2011/2:6
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Primary Sclerosing Cholangitis; Cholangiocarcinoma
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MR/MRCP — MR/MRCP

SUMMARY:
This observational study of a national cohort of 600 Swedish PSC patients include yearly MR/MRCP, biobanking of serum, plasma and blood, followup clinical data (interventions, symptoms, labs, colonoscopy). The aim is to collect a well characterized cohort of PSC patients and provide future possibilities to evaluate biomarkers for prognosis and early cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PSC by MR/MRCP
* Life expectancy >1 year
* Informed consent

Exclusion Criteria:

* Liver transplantation or on the waiting list
* Secondry SC
* Diagnosis of CCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National Swedish cohort of PSC patients followed at 14 hospitals
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
cholangiocarcinoma | 10 yrs f-up
  cholangiocarcinoma
liver transplatation | 10 yrs f-up
  liver transplatation
death | 10 yrs f-up
  death

SECONDARY OUTCOMES:
biliary dysplasia | 10 yrs f-up
  biliary dysplasia

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided